CLINICAL TRIAL: NCT02475928
Title: Zinc Supplementation as Treatment of Dysgeusias in Cirrhotic Patients
Brief Title: Zinc Supplementation in Cirrhotic Patients
Acronym: ZnDCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Clínica Médica Sur (Other)
Responsible Party: Principal Investigator, Norberto Carlos Chavez Taia, Obesity and Digestive Diseases Unit Chief, Fundación Clínica Médica Sur
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Cirrhosis01
Record Dates: First submitted 2015-04-29; First posted 2015-06-19 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Dysgeusia; Liver Cirrhosis
MeSH Terms: conditions — Dysgeusia; Liver Cirrhosis | interventions — gluconic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 100 mg placebo (Placebo Comparator): 100 mg Placebo plus nutritional education
  Interventions: Dietary Supplement: Placebo; Behavioral: Nutritional education
- 100 mg zinc supplement (Experimental): Nutritional education plus 100 mg of zinc gluconate
  Interventions: Dietary Supplement: zinc gluconate; Behavioral: Nutritional education

INTERVENTIONS:
Dietary Supplement: zinc gluconate — Zinc supplementation plus nutritional education
  Arms: 100 mg zinc supplement
Dietary Supplement: Placebo
  Arms: 100 mg placebo
Behavioral: Nutritional education

SUMMARY:
The purpose of this study is to evaluate the effect of zinc supplementation in the treatment for dysgeusia, progression disease and quality of life in patients with liver cirrhosis.

DETAILED DESCRIPTION:
Taste disorders are symptomatologies in patients with cirrhosis, these have a direct effect in modification of food consumption, increasing weight loss, anorexia and malnutrition, which impacts in decompensation rates and mortality.

It has been proposed that zinc deficiency is one of the causes for development of taste disorders. The aim of this study is to describe the presence of taste disorders in patients with cirrhosis and evaluate the effect of zinc supplementation in treatment of taste disorders, and in progression of chronic liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patients by any etiology, with any dysgeusia

Exclusion Criteria:

* Patients with hepatic encephalopathy at the time of dysgeusia evaluation
* Patients with any neurological disease
* Patients with respiratory diseases ath the time of dysgeusia evaluation
* Patients with active alcohol consumption

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-04; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Dysgeusia | Presence of any taste disorder at 6 months
  Evaluation of presence of any taste disorder, according to questionnaires and evaluation of perception and recognition thresholds with ascending molar concentrations of basic tastes.

CONTACTS AND LOCATIONS:
Overall Officials: Norberto C Chávez-Tapia, PhD, Principal Investigator — Medica Sur Clinic & Foundation; Eva Juárez-Hernández, Study Director — Medica Sur Clinic & Foundation
Locations (1):
- Medica Sur Clinic & Foundation, Mexico City, Mexico